CLINICAL TRIAL: NCT03428620
Title: Effect of a Six-week Rehabilitation Program in Conjunction With Thrust Mobilization on Lower Extremity Function in Subjects Reporting Chronic Ankle Instability
Brief Title: Effect of Mobilization in Conjunction With Exercise in Participants With a History of Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenandoah University (Other)
Collaborators: Methodist University, North Carolina (Other)
Responsible Party: Principal Investigator, Cameron Bolton, Assistant Professor Division of Physical Therapy, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 511
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Ankle Sprains
Keywords: Functional Performance; Rehabilitation; Manipulation
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization (Experimental): High Velocity Low Amplitude mobilization group. The three joints that will be manipulated include proximal tibiofibular, the distal tibiofibular, and talocrural joints and will be mobilized the first three sessions prior to the participants performing the exercise protocol.
  Interventions: Other: High Velocity Low Amplitude mobilization; Other: Exercise protocol
- Exercise Protocol (Active Comparator): This exercise regimen is a modified version of the balance training program described by McKeon et al.
  Interventions: Other: Exercise protocol

INTERVENTIONS:
Other: High Velocity Low Amplitude mobilization — Mobilizations will be performed one time at each joint, prior to completing the exercise protocol during the first three treatment sessions.
  Other Names: HVLA; thrust mobilization
  Arms: Mobilization
Other: Exercise protocol — This exercise regimen is a modified version of the balance training program described by McKeon et al.

SUMMARY:
Our purpose is to examine the combined effects of thrust mobilization of the ankle joints in conjunction with a six-week rehabilitation program on functional performance in subjects reporting chronic ankle instability (CAI).

DETAILED DESCRIPTION:
Joint mobilizations are reported to increase range of motion (ROM), postural control and proprioception, and decrease pain in individuals with CAI. However, there is no research supporting the combined effects of thrust mobilization and exercise on function in this population.

Inclusion and exclusion criterion have been established utilizing the International Ankle Consortium guidelines. Using a convenience sampling, participants will be randomized into the exercise only or mobilization (experimental) and exercise group. Both groups will undergo 12 supervised training sessions across a six-week period. The mobilization (experimental) group will also receive high-velocity-low-amplitude (HVLA) thrust mobilizations at the talocrural, proximal, and distal tibiofibular joints prior to the first three treatment sessions.

An examiner, who is blinded to involved limb and group allocation, will perform a baseline and six-week follow-up examination of joint mobility, range of motion, and functional performance. The participants will complete subjective outcome measures at baseline, 2 weeks, 4 weeks, and 6 weeks including the Foot and Ankle Ability Measurement (FAAM), FAAM-Sport, Ankle Joint Functional Assessment Tool (AJFAT), and the Cumberland Ankle Instability Tool (CAIT). Participants will also complete baseline and six-week follow up assessments of the figure-of-8 hop test, side hop test, and three directions of the Star Excursion Balance test (SEBT).

The exercise protocol is a modified version of the balance training program described by McKeon et al. Participants will complete this protocol twice a week for six weeks. Treatment sessions will last approximately 30 minutes. Participants will individually progress on particular exercises if zero errors are observed. In addition, all participants will be given a home exercise program (HEP) to complete every day of the week excluding treatment days.

The mobilization (experimental) group will receive HVLA thrust mobilizations at the three joints stated above for the first three sessions prior to completing the exercise protocol. Each mobilization will be performed one time at each joint. The order of joint mobilizations will be randomized prior to administering.

Data analysis will be performed using International Business Machines Statistical Package for the Social Sciences (SPSS). Alpha level will be set p<0.05. Expecting to utilize separate 2 x 2 repeated measures analysis of variance (ANOVA) to assess changes in the FAAM, FAAM-Sport, AJFAT, CAIT, figure-of-8 hop test, side hop test, and three directions of the SEBT.

ELIGIBILITY:
As adapted from the position statement from the international ankle consortium.

Inclusion Criteria:

* 18-35 years of age
* A history of at least 1 significant ankle sprain (The initial sprain must have occurred at least 12 months prior to study enrollment, associated with inflammatory symptoms (pain, swelling, etc), created at least 1 interrupted day of desired physical activity)
* The most recent injury must have occurred more than 3 months prior to study enrollment.
* A history of the previously injured ankle joint "giving way" and/or recurrent sprain and/or "feelings of instability."
* Cumberland Ankle Instability Tool (CAIT) < 24
* Foot and Ankle Ability Measure (FAAM)42: ADL scale < 90%, Sport scale < 80%

Exclusion Criteria:

* A history of previous surgeries to the musculoskeletal structures (ie, bones, joint structures, nerves) in either limb of the lower extremity.
* A history of a fracture in either limb of the lower extremity requiring realignment
* Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months, which impacted joint integrity and function (ie, sprains, fractures) resulting in at least 1 interrupted day of desired physical activity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in baseline Figure-of-8 hop test at 6 weeks. | Baseline and 6 weeks
  The participant begins the test on either side of a demarcated 5-meter distance. While standing on the involved ankle, the participant is instructed to "hop on one foot, as fast as you can," twice around the figure 8. Two trials will be performed with the fastest time being recorded.
Change in baseline Side hop test at 6 weeks | Baseline and 6 weeks
  The participant stands on the involved limb on either side of two lines that are 30 cm apart. They are then instructed to "hop on one foot, as fast as you can," laterally and then back to the starting position. This is counted as two repetitions and 10 repetitions are performed. If the participant lands on or between the lines, this repetition does not count and they continue until 10 good repetitions are completed. Participants perform two trials and the fastest time is recorded.
Change in baseline Star Excursion Balance Test (SEBT) at 6 weeks | Baseline and 6 weeks
  Each participant is asked to maintain single-limb stance, with hands on their hips, while reaching in anterior, posteromedial, and posterolateral directions.
Change in baseline Foot and Ankle Ability Measure (FAAM)- Activities of Daily Living (ADL) Subscale at 6 weeks | Baseline and 6 weeks
  The FAAM- ADL is a 21-item tool that is designed to assess functional limitations related to foot and ankle conditions. Each item is scored on a Likert scale; 0 (unable to do) to 4 (no difficulty) and has total point value of 84 points, reported as a percent value.
Change in baseline Foot and Ankle Ability Measure (FAAM)- Sport subscale at 6 weeks | Baseline and 6 weeks
  The FAAM- Sport is a 7-item tool that is a sub-scale of the FAAM. Each item is scored on a Likert scale; 0 (unable to do) to 4 (no difficulty) with a total point value of 28 points, reported as a percent value.
Change in baseline Ankle Joint Functional Assessment Tool (AJFAT) at 6 weeks | Baseline and 6 weeks
  12-item tool that rates the participant's overall perceived level of function. Each item is assigned a point value from 0 (much less than other ankle) to 4 (much more than other ankle) with a possible total value of 48 points.
Change in baseline Cumberland Ankle Instability Tool (CAIT) at 6 weeks. | Baseline and 6 weeks
  9-item questionnaire that helps discriminate and measure the severity of functional ankle instability.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron J Bolton, DPT, Principal Investigator — Shenandoah University; Sheri Hale, PhD, PT, Principal Investigator — Shenandoah University
Locations (2):
- United States (2):
  - Methodist University, Fayetteville, North Carolina
  - Shenandoah University, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gribble PA, Delahunt E, Bleakley CM, Caulfield B, Docherty CL, Fong DT, Fourchet F, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino W, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Athl Train. 2014 Jan-Feb;49(1):121-7. doi: 10.4085/1062-6050-49.1.14. Epub 2013 Dec 30. PMID 24377963
- [Background] McKeon PO, Ingersoll CD, Kerrigan DC, Saliba E, Bennett BC, Hertel J. Balance training improves function and postural control in those with chronic ankle instability. Med Sci Sports Exerc. 2008 Oct;40(10):1810-9. doi: 10.1249/MSS.0b013e31817e0f92. PMID 18799992
- [Background] Hale SA, Hertel J, Olmsted-Kramer LC. The effect of a 4-week comprehensive rehabilitation program on postural control and lower extremity function in individuals with chronic ankle instability. J Orthop Sports Phys Ther. 2007 Jun;37(6):303-11. doi: 10.2519/jospt.2007.2322. PMID 17612356
- [Background] Beazell JR, Grindstaff TL, Sauer LD, Magrum EM, Ingersoll CD, Hertel J. Effects of a proximal or distal tibiofibular joint manipulation on ankle range of motion and functional outcomes in individuals with chronic ankle instability. J Orthop Sports Phys Ther. 2012 Feb;42(2):125-34. doi: 10.2519/jospt.2012.3729. Epub 2012 Feb 1. PMID 22333567